CLINICAL TRIAL: NCT04755478
Title: Ultrasound Assessment of Aeration Changes After Lung Lobectomy: a Pilot Study
Brief Title: LUS to Assess Lung Injury After Lung Lobectomy
Acronym: OPEN THORUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Ana Broseta Lleó, Principal Investigator, Hospital General Universitario de Valencia
Other Study IDs: OPEN THORUS
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Lung Neoplasm; Adult ALL; Lung Injury; Lung Inflammation; Lung Ischemia/Hypoxia; Postoperative Complications; Postoperative Respiratory Complication; Lung Cancer; Thoracic
Keywords: thoracic surgery; lung ultrasound; cytokines blood; lung injury; postoperative complications
MeSH Terms: conditions — Lung Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lung Injury; Pneumonia; Hypoxia; Postoperative Complications | interventions — Thoracotomy; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung lobectomy via open thoracotomy: participants scheduled for lung lobectomy via open thoracotomy
  Interventions: Procedure: Thoracotomy
- Lung lobectomy via VATS: participants scheduled for lung lobectomy via video-assisted thoracoscopic surgery
  Interventions: Procedure: VATS

INTERVENTIONS:
Procedure: Thoracotomy — Participants will undergo lobectomy via open thoracotomy at the discretion of the surgical team.
  Groups: Lung lobectomy via open thoracotomy
Procedure: VATS — Participants will undergo lobectomy via VATS at the discretion of the surgical team.
  Groups: Lung lobectomy via VATS

SUMMARY:
The purpose of the study is to assess whether lung ultrasound is able to detect lung injury after lung resection surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPC) are common after lung resection surgery, with an incidence that ranges between 11-32%. As PPC are associated with worse outcomes, many studies aim to find predictors that identify high risk patients and prompt specific interventions and/or monitoring and hence, improve outcomes. PPC result from lung injury inherent to lung resection surgery. Lung aeration changes seen with lung ultrasound (LUS) could detect lung injury and thus, identify patients at high risk of PPC. The underlying mechanisms of lung injury are different in the dependent and non-dependent lung; oxidative stress in both lungs, lung injury associated with one-lung ventilation in the dependent lung and ischemia/reperfusion or surgical manipulation in the non-dependent lung. LUS evaluates the dependent and non-dependent lung separately and so it can be valuable in understanding the characteristics and intensity of lung injury in each lung specifically.

This is a prospective, single-centre, observational study in which 30 consecutive participants with non-small cell lung cancer scheduled for lobectomy will be recruited. Participants will be divided in two groups depending on the surgical approach. First group will be lobectomy via thoracotomy. Second group will be lobectomy via VATS. Participants will be recruited consecutively until there are 15 patients in each group. LUS will be performed in each participant's operated and non-operated lung at three predefined time points: before surgery, after extubation and 24 h after surgery. Each hemithorax will be divided into 6 areas: anterior, lateral and posterior, separated by the anterior and posterior axillary lines, each divided into upper and lower zones. For each echographic examination, cineloops of the most pathological findings in each area will be stored and analysed offline by two independent and blinded anaesthesiologists. From these, a semiquantitative score, the modified lung ultrasound score (mLUSS), will be calculated for each hemithorax to assess lung aeration at each time point. The level of agreement for mLUSS will be tested. At the same predefined time points blood plasma samples will be collected, flash-frozen and stored in order to measure levels of the inflammatory mediators IL-6, IL-10 and TNFα.

The investigators hypothesise that LUS can detect lung injury after lung resection surgery. The primary objective of the study is to assess changes in lung aeration after lung resection with mLUSS. Secondary objectives are, first, to describe LUS findings after lung resection surgery, second, to assess the ability of mLUSS to detect oxygenation changes after lung resection and third, to compare the behaviour of inflammatory mediators in plasma with mLUSS changes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* ASA I-III
* Non-small cell lung neoplasm
* Elective lung lobectomy
* Under one-lung ventilation

Exclusion Criteria:

* Pregnancy
* Respiratory tract infection the previous month
* Diagnosed pulmonary fibrosis
* Predicted FEV < 40%
* Surgery that includes resection of the thoracic wall or the diaphragm
* Neoplasm metastasis
* Obesity class II or more (BMI ≥ 35 kg/m^2)
* Risk of malnutrition CONUT > 1
* Hemoglobin < 10 g/dl
* Chronic kidney failure: glomerular filtration < 60 ml/min/m^2, nephrectomy, kidney transplantation
* Treatment with corticosteroids or immunosuppressive agents 3 months before surgery
* Transfusion of blood products during the previous 10 days
* Heart failure (New York Heart Association Functional Class 3 or 4) during the week before surgery.
* Heart valve diseases over stage B of the American College of Cardiology/American
* Heart Association Task Force on Practice Guidelines 2014
* Diastolic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients assigned to a tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in mLUSS after lung resection. | preoperative vs immediate postoperative period vs 24 hours after surgery.
  The modified lung ultrasound score (mLUSS) ranges 0-36; the higher the score, the less aeration (worse).

SECONDARY OUTCOMES:
LUS feasibility in the dependent and non-dependent lung. | Preoperative vs immediate postoperative period vs 24 hours after surgery.
  Percetage of patients in which ultrasound examination is feasible. There is no important surgical emphysema and/or the dressings or chest tubes do not preclude the feasibility of the examination.
Changes in oxygenation (PAFI) after lung resection. | Preoperative vs immediate postoperative vs 24 hours after surgery.
  PAFI is the ratio between paO2 and fraction of inspired oxygen; the lower, the worse.
Changes in plasma cytokine IL-6 after lung resection. | Preoperative vs immediate postoperative vs 24 hours after surgery.
Changes in plasma cytokine IL-10 after lung resection. | Preoperative vs immediate postoperative vs 24 hours after surgery.
Changes in plasma TNFα after lung resection. | Preoperative vs immediate postoperative vs 24 hours after surgery.
Changes in blood bone natriuretic peptide (BNP) after lung resection. | Preoperative vs immediate postoperative vs 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Broseta Lleó, Consultant, Principal Investigator — Hospital General Universitario de Valencia
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No